CLINICAL TRIAL: NCT01106014
Title: A Multicenter, Double-blind, Placebo-controlled Phase 3 Study Assessing the Safety and Efficacy of Selexipag on Morbidity and Mortality in Patients With Pulmonary Arterial Hypertension
Brief Title: Selexipag (ACT-293987) in Pulmonary Arterial Hypertension
Acronym: GRIPHON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-065A302
Record Dates: First submitted 2010-04-02; First posted 2010-04-19 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — selexipag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Selexipag is up-titrated from Day 1 to Week 12 to each patient's maximum tolerated dose in the range of 200-1600 µg twice a day (b.i.d.) in 200 µg steps starting with one 200 µg oral tablet on Day 1. From Day 2 onwards, a b.i.d. dose regimen with an interval of approximately 12 hours is followed. If this dose (selexipag 200 μg b.i.d.) is well-tolerated, selexipag is up-titrated with weekly increments of 200 µg. Up-titration is followed by a stable maintenance treatment period from Week 12 onwards, up to Week 26, at the maximum tolerated dose
  Interventions: Drug: Selexipag
- 2 (Placebo Comparator): Matching placebo is administered orally with a dosing interval of approximately12 h. A (mock) up-titration scheme is followed
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selexipag — Selexipag 200 µg tablets
  Other Names: ACT-293987
  Arms: 1
Drug: Placebo — Placebo tablets matching selexipag
  Arms: 2

SUMMARY:
The AC-065A302 (GRIPHON) study is an event-driven Phase 3 study to demonstrate the effect of selexipag on time to first morbidity or mortality event in patients with pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18-75 years old, with symptomatic PAH
* PAH belonging to the following subgroups of the updated Dana Point Clinical Classification Group 1 (Idiopathic, or Heritable, or Drug or toxin induced, or Associated (APAH) with Connective tissue disease, Congenital heart disease with simple systemic-to-pulmonary shunt at least 1 year after surgical repair, or HIV infection)
* Documented hemodynamic diagnosis of PAH by right heart catheterization, performed at any time prior to Screening
* Six minute walk distance (6MWD) between 50 and 450 m at Screening within 2 weeks prior to the Baseline Visit
* Signed informed consent

Exclusion Criteria:

* Patients with pulmonary hypertension (PH) in the Updated Dana Point Classification Groups 2-5, and PAH Group 1 subgroups that are not covered by the inclusion criteria
* Patients who have received prostacyclin or its analogs within 1 month before Baseline Visit, or are scheduled to receive any of these compounds during the trial
* Patients with moderate or severe obstructive lung disease
* Patients with moderate or severe restrictive lung disease
* Patients with moderate or severe hepatic impairment (Child-Pugh B and C)
* Patients with documented left ventricular dysfunction
* Patients with severe renal insufficiency
* Patients with BMI <18.5 Kg/m2
* Patients who are receiving or have been receiving any investigational drugs within 1 month before the Baseline Visit
* Acute or chronic impairment (other than dyspnea), limiting the ability to comply with study requirements, in particular with 6MWT
* Recently conducted or planned cardio-pulmonary rehabilitation program based on exercise training
* Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements
* Life expectancy less than 12 months
* Females who are lactating or pregnant or plan to become pregnant during the study
* Known hypersensitivity to any of the excipients of the drug formulations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1156 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aline Frey, Study Director — Actelion
Locations (182):
- United States (43):
  - University of South Alabama, Mobile, Alabama
  - The University of Arizona, Clinical and Translational Science (CATS) Research Center, Tucson, Arizona
  - University of California San Diego Medical Center (La Jolla), La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - GLVA Healthcare Center, Los Angeles, California
  - University of California, Davis, UC Davis Medical Center, Sacramento, California
  - LIU Center for Pulmonary Hypertension, Torrance, California
  - Lung Health & Sleep Emhancement Center, LLC, Newark, Delaware
  - Emory University School of Medicine, Division of Pulmonary, Allergy and Critical Care Medicine, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - Georgia Clinical Research, Austell, Georgia
  - Clarian North Hospital, Carmel, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - LSU Health Science Center - New Orleans, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital - Pulmonary Critical Care Unit, Boston, Massachusetts
  - Massachusetts General Hospital-Pulmonary Critical Care Unit, Boston, Massachusetts
  - Boston University School of Medicine / Boston University Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Beaumont Hospital, Troy, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Newark Beth Isreal Medical Center-Department of Pulmonary Medicine, Newark, New Jersey
  - Columbia University Medical Center, Pediatric Cardiology, New York, New York
  - Montefiore Medical Center, Weiler Division, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Pulmonary Associates, PC, Portland, Oregon
  - Central Bucks Specialists, Doylestown, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas-Houston Health Center Department of Pulmonary & Critical Care, Houston, Texas
  - University of Wisconsin Hospital-Department of Medicine, Madison, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert Hospital - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (6):
  - Centro de Investigacion y Prevencion Cardiovascular (CIPREC), Buenos Aires
  - Sanatorio Otamendi y Miroli S.A., Buenos Aires
  - Hospital Britanico-Pneumology, Buenos Aires
  - Sanatorio San Jose, Buenos Aires
  - Instituto De Cardiologia de Corrientes, Corrientes
  - Hospital Privado Centro Medico de Cordoba S.A., Córdoba
- Australia (9):
  - St. Vincent's Hospital / Heart and Lung Transplant Unit, Darlinghurst, New South Wales
  - Prince Charles Hospital Lung Transplant, Thoracic Department, Chermside, Queensland
  - Royal Adelaide Hospital, Cardiovascular Investigation Unit (CVIU), Adelaide, South Australia
  - Flinders Medical Centre, Pulmonary Hypertension, c/- Cardiology, Bedford Park, South Australia
  - St Vincent's Hospital, Fitzroy, Victoria
  - Royal Hobart Hospital, Centre for Clinical Research, Hobart
  - John Hunter Hospital Autoimmune Resource and Research Centre, New Lambton
  - Royal Melbourne Hospital, Department of Respiratory and Sleep Medicine, Parkville
  - Royal Perth Hospital, Perth
- Austria (2):
  - Medizinische Universität Graz, Graz
  - Medical University of Vienna and AKH Cardiology, Vienna
- Belarus (3):
  - The Republican Scientific-Practical Center "Cardiology", Minsk
  - Minsk City Hospital No. 9, Minsk
  - Minsk Regional Clinical Hospital of the Red Banner of Labour, Minsk
- Belgium (2):
  - Ulb Erasme, Cardiology, Brussels
  - University Hospital Gasthuisberg - Pneumologie, Leuven
- Canada (7):
  - University of Alberta Hospital - Children's Centre, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Hopital General Juif (Jewish General Hospital), Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
- Chile (3):
  - Instituto Nacional del Torax Teaching Dept, Santiago
  - Clinica Tabancura- Cardiology Unit, Santiago
  - Pontificia Universidad Catolica de Chile-Departmento De Enfermedades Cardiovasculares, Santiago
- China (7):
  - Peking Union Medical College Hospital, Rheumatology Department, Beijing
  - Cardiovascular Institute & Fuwai Hospital-Pulmonary Vascular Center, Beijing
  - Beijing Shijitan Hospital, Beijing
  - Guangdong General Hospital, Cardiology Department, Guangzhou
  - Renji Hospital, Rheumatology Department, Shanghai
  - Renji Hospital, Cardiology Department, Shanghai
  - Shanghai Pulmonary Hospital, Department of Pulmonary Circulation, Shanghai
- Colombia (2):
  - Fundacion Cardio Infantil, Bogotá
  - Fundacion Clinica Shaio, Bogotá
- Gen Faculty Hosp Prague Cardiology Clin, Prague, Czechia
- Denmark (2):
  - Aarhus University Hospital , Cardiology, Aarhus
  - Rigshospitalet, Hjertemedicinsk klinik - Cardiology, Copenhagen
- France (6):
  - Hosp Pradel Lyon - Dpt Pneumology, Bron
  - Hosp Cote de Nacre - Dpt Pneumology, Caen
  - Hosp A. Beclere - Dept Pulmo & Resp Intensive Care, Clamart
  - Hosp Huriez - Dpt Internal Medecine, Lille
  - Hosp Civil - Dpt Pneumology, Strasbourg
  - Hosp Larrey - Dpt Pneumology, Toulouse
- Germany (10):
  - DRK Kliniken Köpenick, Berlin
  - "Universitätsklinikum Köln Herzzentrum / Klinik III für Innere Medizin (Kardiologie, Pneumologie, Angiologie und Intensivmedizin)", Cologne
  - Universitätsklinikum Carl Gustav Carus, Medizinische Klinik1-Pneumologie/MK1-A13, Dresden
  - "Justus-Liebig-Universität Gießen Zentrum für Innere Medizin Medizinische Klinik II", Giessen
  - Universität Greifswald / Klinik für Innere Medizin B, Greifswald
  - Medizinische Hochschule Hannover / Klinik für Pneumologie, Hanover
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Praxis für Pneumologie und Allergologie, Leipzig
  - Klinik Löwenstein gGmbH, Medizinische Klinik 1, Pneumologie - Kardiologie, Löwenstein
  - Universitätsklinkum Regensburg / Innere Medizin II, Regensburg
- Onasseio Cardiosurgical Hospital, Athens, Greece
- Hungary (5):
  - "Gottsegen György Országos Kardiológiai Intézet, Felnőtt kardiológiai osztály", Budapest
  - "Semmelweis Egyetem, Pulmonológiai Klinika", Budapest
  - Egészségügyi Járóbeteg Központ Kardiológiai Intézete - Debrecen, Debrecen
  - "Pécsi Tudományegyetem Klinikai Központ,, Pécs
  - "Szegedi Tudományegyetem ÁOK Szent-Györgyi Albert Klinikai Központ, II. sz. Belgyógyászati klinika és Kardiológiai központ", Szeged
- India (5):
  - Sanjivani Hospitals - Department of Cardiology, Ahmedabad
  - Apollo Hospitals, Chennai, Chennai
  - Frontier Lifeline Hospitals, Dr KM Cherian Heart Foundation, Chennai, Chennai
  - CARE Hospitals Nampally, Cardiology Dep. Hyderabad, Hyderabad
  - Apollo Indraprastha Hospitals, New Delhi
- Mater Miscordiae University Hospital, Dublin, Ireland
- Israel (5):
  - Carmel Medical Center, Pulmonary Unit, Haifa
  - Pulmonology Institute, Hadassah University Hospital at Ein Karem, Jerusalem
  - Rabin Medical Centre - Pulmonology, Petach Tikvah
  - Kaplan Medical - Pulmonary Institute, Rehovot
  - The Chaim Sheba Med Ctr -Pulmonology, Tel Litwinsky
- Italy (3):
  - Policlinico S. Orsola-Malpighi - Dipartimento Cardio-Toraco-Vascolare, Bologna
  - Seconda Università Degli Studi di Napoli - Azienda Universitaria Policlinico - Dipartimento Assistenziale di medicina Generale, Angiologia, Endocrinologia, Epatogastroenterologia e Reumatologia - Unità Operativa di Reumatologia, Napoli
  - ISMETT - Istituto Mediterraneo Trapianti e Terapie ad Alta Specializzazione - Dipartimento di Medicina - Divisione di Pneumologia, Palermo
- Institut Jantung Negara (National Heart Institute), Kuala Lumpur, Malaysia
- Mexico (2):
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubrian, Mexico City
  - Instituto Nacional de Cardiologia (INC) Ignacio Chavez, Mexico City
- Netherlands (4):
  - VU Medisch Centrum / Afdeling longziekten, secretariaat 4A 48, Amsterdam
  - Academisch Ziekenhuis Maastricht / Department of Pulmonary Diseases, Maastricht
  - St. Antonius Ziekenhuis afdeling Longziekten, Nieuwegein
  - Erasmus Medisch Centrum Rotterdam afdeling longziekten, Rotterdam
- Peru (2):
  - Hospital Nacional Edgardo Rebagliati / Unidad de Investigacion Cardiologia 2, Lima
  - Instituto de Enfermedades Respiratorias Clinica San Gabriel, Lima
- Poland (4):
  - "Uniwersyteckie Centrum Kliniczne II Klinika Kardiologii i Elektroterapii Serca", Gdansk
  - "Instytut Kardiologii Collegium Medium UJ Krakowski Szpital Specjalistyczny im Jana Pawła II Klinika Chorób Serca i Naczyń", Krakow
  - "Wojewódzki Specjalistyczny Szpital im. dr Władysława Biegańskiego Oddział Kardiologiczny, II Katedra i Klinika Kardiologii UM", Lodz
  - "Instytut Gruźlicy i Chorób Płuc Klinika Chorób Wewnętrznych Klatki Piersiowej", Warsaw
- Romania (2):
  - "Institutul de Pneumologie "Marius Nasta", I. Clinica de Pneumoftiziologie", Bucharest
  - "Spitalul Clinic de Pneumoftiziologie Iasi Sectia Clinica I de Pneumoftiziologie", Iași
- Russia (10):
  - Municipal Medical Institution City Hospital #5, Barnaul
  - Kemerovo Cardiology Dispensary / Kemerovo Regional Hospital, Kemerovo
  - Scientific Research Institute of Pulmonology of the Federal Medical and Biological Agency of Russia, Moscow
  - State Institution, "Institute fo Rheumatology of RAMS", Moscow
  - The Institution of the Clinical Cardiology named after A. L. Myaskinov, Moscow
  - Limited liability company, Consultative diagnostic centre Healthy Joints, Novosibirsk
  - V. A. Almazov Institute of Cardiology, Russian Ministry of Healthcare and Social Development / Medical Treatment and Rehabilitation Complex, Saint Petersburg
  - Cardiology Scientific Research Institute of Tomsk Scientific Center of RAMs, Siberian Branch / Cardiovascular Surgery Department, Tomsk
  - Tomsk Regional Clinical Hospital/ Pulmonology Unit, Tomsk
  - Regional Clinical Hospital # 1, Yekaterinburg
- Serbia (2):
  - "Klinički Centar Srbije, Klinika za pulmologiju", Belgrade
  - "Kliničko-bolnički centar Zemun, Kardiološko odeljenje", Belgrade
- National Heart Centre (NHC) Singapore, Singapore, Singapore
- Národný ústav srdcových a cievnych chorôb, a.s. - NÚSCH a.s., Bratislava, Slovakia
- South Korea (5):
  - Gil Medical Centre, Incheon
  - Seoul Nathional University Hospital, Seoul
  - Yonsei University Health System Dept of Cardiology, Seoul
  - Samsung Medical Center, Division of Cardiology, Seoul
  - "The Catholic University of Korea, Seoul St. Mary's Hospital Department of Cardiology", Seoul
- Spain (3):
  - Hosp Vall D'Hebron - Barcelona - Pneumology, Barcelona
  - Clinic-Barcelona, Barcelona
  - Hospital 12 Octubre, Madrid
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset, Kardiologi, Gothenburg
  - Linköping University Hospital, Cardiology, Linköping
  - Umeå University Hospital, Cardiology (Umeå), Umeå
  - Uppsala Akademiska Sjukhuset, Kardiologkliniken 50F, Uppsala
- Switzerland (4):
  - University Hospital Basel Division of Pneumology, Basel
  - Universitätsspital Bern, Clinic for Pneumology (Inselspital), Bern
  - HUG Hôpitaux Universitaires de Genève; Pneumology, PAH, Geneva
  - Kantonsspital St. Gallen Klinik für Pneumologie, Sankt Gallen
- Taiwan (2):
  - Kaohsiung Veterans General Hospital (KVGH), Kaohsiung City
  - National Taiwan University Hospital / Department of Surgery, Taipei
- Srinagarind Hospital, Khon Kaen University, Division of Allergy-Immunology and Rheumatology, Department of Medicine, Khon Kaen, Thailand
- Turkey (Türkiye) (4):
  - Çukurova Üniversitesi Tıp Fakültesi Kardiyoloji Anabilim Dalı, Adana
  - Istanbul Üniversitesi Kardiyoloji Enstitisü, Istanbul
  - Marmara Üniversitesi Tip Fakultesi Kardiyoloji Anabilim Dali, Istanbul
  - Dokuz Eylül Üniversitesi Tıp Fakültesi Kardiyoloji Anabilim Dalı, Izmir
- Ukraine (4):
  - "Dnipropetrovsk State Medical Academy, Municipal Institution ""Dnipropetrovsk Regional Clinic Diagnostic Center"", Dnipropetrovsk
  - Health Care Municipal Institution, City Clinical Hospital #13, Kharkiv
  - Public Institution "F.H. Yanovski Phthisiology and Pulmonology National Institute Under Ukrainian Academy of Medical Sciences", Kyiv
  - Lviv Regional Clinical Hospital, Lviv
- United Kingdom (3):
  - Golden Jubilee - Pulm Vascular Unit, Glasgow
  - Royal Free & Ucms Rheumatology Unit, London
  - Hammersmith, London

REFERENCES:
- [Result] Sitbon O, Channick R, Chin KM, Frey A, Gaine S, Galie N, Ghofrani HA, Hoeper MM, Lang IM, Preiss R, Rubin LJ, Di Scala L, Tapson V, Adzerikho I, Liu J, Moiseeva O, Zeng X, Simonneau G, McLaughlin VV; GRIPHON Investigators. Selexipag for the Treatment of Pulmonary Arterial Hypertension. N Engl J Med. 2015 Dec 24;373(26):2522-33. doi: 10.1056/NEJMoa1503184. PMID 26699168
- [Derived] Benza RL, Chin KM, Gaine S, Galie N, Hoeper MM, Lang IM, McLaughlin VV, Sitbon O, Doad G, Yen J, Tang X, Tapson V. Changes in REVEAL Lite 2 risk status are associated with long-term outcomes in patients with pulmonary arterial hypertension: A post-hoc analysis of the GRIPHON study. J Heart Lung Transplant. 2024 Dec;43(12):1998-2007. doi: 10.1016/j.healun.2024.08.019. Epub 2024 Aug 31. PMID 39222737
- [Derived] Galie N, Gaine S, Channick R, Coghlan JG, Hoeper MM, Lang IM, McLaughlin VV, Lassen C, Rubin LJ, Hsu Schmitz SF, Sitbon O, Tapson VF, Chin KM. Long-Term Survival, Safety and Tolerability with Selexipag in Patients with Pulmonary Arterial Hypertension: Results from GRIPHON and its Open-Label Extension. Adv Ther. 2022 Jan;39(1):796-810. doi: 10.1007/s12325-021-01898-1. Epub 2021 Oct 30. PMID 34727317
- [Derived] Gaine S, Sitbon O, Channick RN, Chin KM, Sauter R, Galie N, Hoeper MM, McLaughlin VV, Preiss R, Rubin LJ, Simonneau G, Tapson V, Ghofrani HA, Lang I. Relationship Between Time From Diagnosis and Morbidity/Mortality in Pulmonary Arterial Hypertension: Results From the Phase III GRIPHON Study. Chest. 2021 Jul;160(1):277-286. doi: 10.1016/j.chest.2021.01.066. Epub 2021 Feb 3. PMID 33545163
- [Derived] Chin KM, Rubin LJ, Channick R, Di Scala L, Gaine S, Galie N, Ghofrani HA, Hoeper MM, Lang IM, McLaughlin VV, Preiss R, Simonneau G, Sitbon O, Tapson VF. Association of N-Terminal Pro Brain Natriuretic Peptide and Long-Term Outcome in Patients With Pulmonary Arterial Hypertension. Circulation. 2019 May 21;139(21):2440-2450. doi: 10.1161/CIRCULATIONAHA.118.039360. PMID 30982349
- [Derived] McLaughlin VV, Hoeper MM, Channick RN, Chin KM, Delcroix M, Gaine S, Ghofrani HA, Jansa P, Lang IM, Mehta S, Pulido T, Sastry BKS, Simonneau G, Sitbon O, Souza R, Torbicki A, Tapson VF, Perchenet L, Preiss R, Verweij P, Rubin LJ, Galie N. Pulmonary Arterial Hypertension-Related Morbidity Is Prognostic for Mortality. J Am Coll Cardiol. 2018 Feb 20;71(7):752-763. doi: 10.1016/j.jacc.2017.12.010. PMID 29447737
- [Derived] Coghlan JG, Channick R, Chin K, Di Scala L, Galie N, Ghofrani HA, Hoeper MM, Lang IM, McLaughlin V, Preiss R, Rubin LJ, Simonneau G, Sitbon O, Tapson VF, Gaine S. Targeting the Prostacyclin Pathway with Selexipag in Patients with Pulmonary Arterial Hypertension Receiving Double Combination Therapy: Insights from the Randomized Controlled GRIPHON Study. Am J Cardiovasc Drugs. 2018 Feb;18(1):37-47. doi: 10.1007/s40256-017-0262-z. PMID 29307087
- [Derived] Gaine S, Chin K, Coghlan G, Channick R, Di Scala L, Galie N, Ghofrani HA, Lang IM, McLaughlin V, Preiss R, Rubin LJ, Simonneau G, Sitbon O, Tapson VF, Hoeper MM. Selexipag for the treatment of connective tissue disease-associated pulmonary arterial hypertension. Eur Respir J. 2017 Aug 17;50(2):1602493. doi: 10.1183/13993003.02493-2016. Print 2017 Aug. PMID 28818881
- [Derived] Krause A, Machacek M, Lott D, Hurst N, Bruderer S, Dingemanse J. Population Modeling of Selexipag Pharmacokinetics and Clinical Response Parameters in Patients With Pulmonary Arterial Hypertension. CPT Pharmacometrics Syst Pharmacol. 2017 Jul;6(7):477-485. doi: 10.1002/psp4.12202. Epub 2017 May 27. PMID 28556581
- [Derived] Skoro-Sajer N, Lang IM. Selexipag for the treatment of pulmonary arterial hypertension. Expert Opin Pharmacother. 2014 Feb;15(3):429-36. doi: 10.1517/14656566.2014.876007. Epub 2014 Jan 7. PMID 24392948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1351 patients were screened from 181 sites in 39 countries worldwide. Of these, 1156 were randomized
Pre-assignment Details: Screening assessments were performed up to a maximum of 28 days before baseline
Groups:
- SELEXIPAG: During the 12-week titration phase, treatment was initiated at 200 μg twice daily (b.i.d.) and up-titrated weekly in 200 μg b.i.d. increments to the maximum tolerated dose (MTD) for each individual patient but not above 1600 μg b.i.d. At Week 12, patients continued the treatment at their individual MTD up to Week 26. Thereafter the dose could be up-titrated at scheduled visits if needed for patients receiving a dose < 1600 μg b.i.d. The dose could be decreased at any time in case of tolerability issues.
- PLACEBO: Matching placebo was administered orally following the same administration schedule as described for selexipag
Period: Overall Study
Arm/Group | SELEXIPAG | PLACEBO
Started | 574 | 582
Completed | 289 | 252
Not Completed | 285 | 330
Not completed — Morbidity or Mortality primary endpoint | 155 | 242
Not completed — Adverse Event | 78 | 42
Not completed — Withdrawal by Subject | 43 | 37
Not completed — Administrative reason | 7 | 6
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selexipag | Placebo | Total
Number analyzed (Participants) | 574 | 582 | 1156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (15.19) | 47.9 (15.55) | 48.1 (15.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 457 | 466 | 923
  Male | 117 | 116 | 233
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasion / White | 376 | 375 | 751
  Asian | 125 | 120 | 245
  Hispanic | 51 | 63 | 114
  Black | 13 | 14 | 27
  Other | 9 | 10 | 19
Region of Enrollment [Number; unit: Participants]
  Western Europe & Australia | 161 | 160 | 321
  Eastern Europe | 149 | 155 | 304
  Asia | 115 | 113 | 228
  North America | 95 | 98 | 193
  Latin America | 54 | 56 | 110
PAH etiology [Number; unit: Participants] — Number of patients in each PAH etiology category
  Participants
    Idiopathic | 312 | 337 | 649
    Heritable | 13 | 13 | 26
    Associated with connective tissue disease | 167 | 167 | 334
    Assoc. with corrected (>=12Mo) congenital shunts | 60 | 50 | 110
    Associated with drug or toxin exposure | 17 | 10 | 27
    Associated with HIV infection | 5 | 5 | 10
Modified NYHA/WHO Functional class (FC) [Number; unit: Participants] — Number of patients in each NYHA/WHO Functional class (FC) at screening. The WHO FC ranges from I to IV, with higher ranges indicating more severe functional restrictions
  Participants
    FC I | 4 | 5 | 9
    FC II | 274 | 255 | 529
    FC III | 293 | 314 | 607
    FC IV | 3 | 8 | 11
PAH medications at baseline [Number; unit: Participants] — Number of patients receiving PAH background medication at the time of study drug start
  Participants
    None | 112 | 124 | 236
    Endothelin Receptor Agonists (ERA) | 94 | 76 | 170
    Phosphodiesterase type 5 inhibitors (PDE5-I) | 189 | 185 | 374
    ERA and PDE5I in combination | 179 | 197 | 376
Time since PAH diagnosis [Median (Full Range); unit: Years] | 0.9 [0.0 to 37.3] | 1.1 [0.0 to 38.9] | 1.0 [0.0 to 38.9]
6-minute walk distance (6MWD) at baseline [Median (Full Range); unit: Meters] | 376 [90 to 482] | 369 [50 to 515] | 372 [50 to 515]

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to the First Morbidity Event or Death (All Causes) up to 7 Days After the Last Study Drug Intake
Description: Time from randomization to the first occurrence of a morbidity event or death (all causes) was analyzed with the Kaplan-Meier method (event-free KM estimates at different time points).
  Morbidity event was defined as any of the following events confirmed by the Critical Event committee:
  * Hospitalization for worsening of pulmonary arterial hypertension (PAH),
  * Worsening of PAH resulting in need for lung transplantation or balloon atrial septostomy,
  * Initiation of parenteral prostanoid therapy or chronic oxygen therapy due to worsening of PAH,
  * Disease progression which was defined by a decrease in 6-minute walk distance from baseline (>=15%, confirmed by a 2nd test on a different day) combined with worsening of WHO FC for patients belonging to WHO FC II/III at baseline, or combined with the need for additional PAH-specific therapy for patients belonging to WHO FC III/IV at baseline.
  Note: The number of patients at risk decreased over time but this cannot be captured below
Time Frame: Up to 7 days after end of double-blind treatment (maximum: 4.3 years)
Population: The primary endpoint was analyzed using the full analysis set, which includes all randomized patients evaluated according to the study drug to which they have been randomized (intention-to treat analysis set).
Measure: Number (95% Confidence Interval); unit: Percentage of patients free of events
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 574 | 582
Percentage of patients free of events
  KM estimate at Month 6 | 91.2 [88.5 to 93.4] | 81.7 [78.2 to 84.7]
  KM estimate at Month 12 | 83.1 [79.5 to 86.1] | 70.6 [66.6 to 74.3]
  KM estimate at Month 18 | 75.5 [71.2 to 79.2] | 61.3 [56.8 to 65.5]
  KM estimate at Month 24 | 67.9 [63.0 to 72.4] | 53.9 [49.0 to 58.5]
  KM estimate at Month 30 | 61.9 [56.3 to 66.9] | 49.3 [44.2 to 54.3]
  KM estimate at Month 36 | 58.2 [51.7 to 64.1] | 41.7 [35.2 to 48.0]
Statistical Analysis 1: Comparison: Selexipag vs Placebo; The primary analysis was performed on the Full Analysis Set by a one-sided unstratified log-rank test; Test type: Superiority or Other; p < 0.0001, Log Rank — one-sided p-value; Hazard Ratio (HR) = 0.6, 99% CI 2-sided [0.46 to 0.78]

2. Secondary Outcome: Change From Baseline to Week 26 in 6-minute Walk Distance (6MWD) at Trough
Description: The 6-minute walk distance test (6MWD) is a non-encouraged test performed in a 30 m long flat corridor, where the patient is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. If the patient was used to taking bronchodilators before a walk, he/she was given them 5 to 30 min before the test. Also if the patient was on chronic oxygen therapy, oxygen was given at their standard rate during the test. Absolute change from baseline to Week 26 in 6MWD was measured at trough, i.e., either on the next day after the last study drug administration or at least 12 hours after study drug administration if on the same day.
Time Frame: Week 26
Population: Full analysis set
Measure: Median (Full Range); unit: Meters
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 574 | 582
Meters
  6MWD at baseline - Overall | 376 [90 to 482] | 369 [50 to 515]
  6MWD at Week 26- Overall | 370 [0 to 617] | 346 [0 to 650]
  6MWD Change from baseline at Week 26 | 4 [-448 to 260] | -9 [-438 to 262]
Statistical Analysis 1: Comparison: Selexipag vs Placebo; Non-parametric ANCOVA with 6MWD as covariate at baseline. Missing values were imputed based on the following imputation rules: 1) if patient was unable to walk at week 26, 0 meter was imputed, 2) if rule 1 did not apply, the second lowest observed 6MWD value (10 meters) at Week 26 was imputed. Missing values were imputed for 21.6% of the subjects; Test type: Superiority or Other; p = 0.0027, ANCOVA — One-sided p-value of the nonparametric ANCOVA, adjusted for 6-minute walk distance at baseline; Median Difference (Final Values) = 12, 99% CI 2-sided [1 to 24] — Point estimate and 2-sided 99% CI for location shift using the HodgesLehmann method

3. Secondary Outcome: Absence of Worsening From Baseline to Week 26 in Modified NYHA/WHO Functional Class (WHO FC)
Time Frame: Week 26
Population: Full analysis set. Patients with WHO FC IV at baseline were excluded from this analysis as they could not shift to a worse category
Measure: Number; unit: Percentage of patients
Arm/Group | Selexipag | Placebo
Number analyzed (Participants) | 571 | 574
Percentage of patients | 77.8 | 74.9
Statistical Analysis 1: Comparison: Selexipag vs Placebo; Test type: Non-Inferiority or Equivalence — It was assumed that the probabilities for absence of worsening in WHO FC at Week 26 were the same for both treatment groups; p = 0.2843, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test stratified by WHO FC at baseline. For patients with missing NYHA/WHO FC at Week 26, the NYHA/WHO FC is considered as having worsened from baseline at Week 26. Missing values were imputed for 18.3% of subjects; Odds Ratio, log = 1.161, 99% CI 2-sided [0.811 to 1.664]

ADVERSE EVENTS:
Time Frame: From baseline up to up to 7 days after end of treatment (EOT)
Description: Median duration of exposure to study drug was 70.7 weeks (range: 0.3-216.7 weeks) in the selexipag group and 63.7 weeks (range: 0.7-192.0 weeks) in the placebo group
Groups:
- Selexipag: This group includes patients who received at least one dose of selexipag. One subject who was randomized to placebo received a single dose of 8 tablets of selexipag due to an error in the dispensation of the medication bottle. Therefore, this patient was assigned to the selexipag group in the safety analysis set.
- Placebo: This group includes patients who received at least one dose of placebo. Four patients who were randomized to placebo never received the drugs and another patient received selexipag by mistake (see Selexipag group for more details). Therefore, these patients were excluded from the placebo group in the safety analysis set.
Arm/Group | Selexipag | Placebo
Serious Adverse Events (participants affected / at risk) | 252/575 | 272/577
Other Adverse Events (participants affected / at risk) | 544/575 | 486/577
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selexipag (N=575) | Placebo (N=577)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (6) | 4 (4)
ABSCESS INTESTINAL (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1)
ABSCESS ORAL (Infections and infestations) | 0 (0) | 1 (1)
ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1)
ACUTE LUNG INJURY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ACUTE RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 2 (2) | 5 (5)
AGEUSIA (Nervous system disorders) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (1)
ALCOHOLISM (Psychiatric disorders) | 0 (0) | 1 (3)
ANAEMIA (Blood and lymphatic system disorders) | 5 (7) | 3 (5)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (2)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 1 (2)
ANURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
APHASIA (Nervous system disorders) | 0 (0) | 1 (1)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 1 (1)
ASCITES (Gastrointestinal disorders) | 2 (2) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 2 (2) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 7 (9) | 4 (5)
ATRIAL FLUTTER (Cardiac disorders) | 3 (3) | 5 (5)
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1) | 2 (4)
ATRIAL THROMBOSIS (Cardiac disorders) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 (1) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 1 (2)
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 1 (1) | 0 (0)
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
BARIATRIC GASTRIC BALLOON INSERTION (Surgical and medical procedures) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
BASEDOW'S DISEASE (Endocrine disorders) | 1 (1) | 0 (0)
BLADDER NECK SUSPENSION (Surgical and medical procedures) | 0 (0) | 1 (1)
BRADYARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
BRAIN HERNIATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (5)
BREAST CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 6 (7) | 4 (4)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 2 (2) | 4 (4)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 2 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 (2) | 1 (1)
CARDIAC INDEX DECREASED (Investigations) | 1 (1) | 1 (1)
CARDIAC PACEMAKER INSERTION (Surgical and medical procedures) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2 (2) | 2 (2)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 2 (2)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 3 (3) | 1 (1)
CARDIOVERSION (Surgical and medical procedures) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 2 (3) | 0 (0)
CATHETER SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CATHETERISATION CARDIAC (Investigations) | 3 (3) | 1 (1)
CELLULITIS (Infections and infestations) | 3 (4) | 3 (3)
CEREBELLAR SYNDROME (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
CERVICAL CONISATION (Surgical and medical procedures) | 1 (1) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 2 (2) | 0 (0)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 6 (7) | 6 (8)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 (0) | 1 (2)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 2 (2)
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CHOROIDITIS (Eye disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CHRONIC RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 2 (3) | 2 (2)
CIRCULATORY COLLAPSE (Vascular disorders) | 2 (2) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLORECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COR PULMONALE (Cardiac disorders) | 1 (2) | 0 (0)
COR PULMONALE ACUTE (Cardiac disorders) | 0 (0) | 1 (1)
COR PULMONALE CHRONIC (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 (0) | 1 (1)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CREST SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
CRYSTAL ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CYANOSIS (Cardiac disorders) | 0 (0) | 1 (1)
CYSTITIS ESCHERICHIA (Infections and infestations) | 1 (1) | 0 (0)
CYSTOCELE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
DEATH (General disorders) | 1 (1) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (3) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
DEMYELINATION (Nervous system disorders) | 1 (1) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOMYOSITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIABETIC GANGRENE (Infections and infestations) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 3 (3)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
DRUG THERAPY CHANGED (Surgical and medical procedures) | 1 (1) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 13 (17)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTEROCELE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENTEROCOLITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
ERYSIPELAS (Infections and infestations) | 2 (2) | 0 (0)
EXERCISE TOLERANCE DECREASED (General disorders) | 1 (1) | 1 (1)
EXTREMITY NECROSIS (Vascular disorders) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 3 (3) | 6 (8)
FATIGUE (General disorders) | 0 (0) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FLUID RETENTION (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
FLUSHING (Vascular disorders) | 1 (1) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 3 (3) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 3 (3)
GASTROINTESTINAL ANGIODYSPLASIA HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 3 (4)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (2)
GINGIVAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
GLAUCOMA SURGERY (Surgical and medical procedures) | 0 (0) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 2 (2)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0)
HAEMODIALYSIS (Surgical and medical procedures) | 1 (1) | 0 (0)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (7)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC CYST (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC MASS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATITIS C (Infections and infestations) | 0 (0) | 1 (1)
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
HYPOGLYCAEMIC UNCONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
HYPONATRAEMIC SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 3 (3) | 3 (3)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
IMPAIRED HEALING (General disorders) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 2 (3) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (2)
INVESTIGATION (Investigations) | 2 (3) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LIP INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2)
LOCALISED INFECTION (Infections and infestations) | 1 (2) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 4 (4)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
LUNG ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 4 (4) | 2 (2)
LUNG TRANSPLANT (Surgical and medical procedures) | 2 (2) | 1 (1)
LUNG TRANSPLANT REJECTION (Immune system disorders) | 0 (0) | 1 (1)
LUPUS NEPHRITIS (Renal and urinary disorders) | 1 (1) | 0 (0)
LYMPHANGIOSIS CARCINOMATOSA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
LYMPHANGITIS (Infections and infestations) | 1 (1) | 0 (0)
MACULOPATHY (Eye disorders) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MASTECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
MENTAL IMPAIRMENT (Nervous system disorders) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1)
MIXED CONNECTIVE TISSUE DISEASE (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 2 (2)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1)
NASAL SEPTAL OPERATION (Surgical and medical procedures) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NECROTISING COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NODULAR REGENERATIVE HYPERPLASIA (Hepatobiliary disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 3 (4) | 4 (5)
OESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
OLIGURIA (Renal and urinary disorders) | 1 (2) | 0 (0)
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ORTHOPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OXYGEN SATURATION DECREASED (Investigations) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 2 (2) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 0 (0)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
PAROTITIS (Infections and infestations) | 0 (0) | 1 (3)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
PERIPHLEBITIS (Vascular disorders) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 2 (2)
PILONIDAL CYST (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 17 (18) | 25 (30)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
POLYMYOSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
POST HERPETIC NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
POST PROCEDURAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 2 (2) | 1 (1)
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 83 (106) | 127 (183)
PULMONARY ARTERIAL PRESSURE INCREASED (Investigations) | 0 (0) | 1 (1)
PULMONARY ARTERIAL WEDGE PRESSURE INCREASED (Investigations) | 0 (0) | 1 (1)
PULMONARY ARTERY DILATATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY INFARCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY VENO-OCCLUSIVE DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
PYELONEPHRITIS (Infections and infestations) | 2 (2) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 3 (3) | 0 (0)
PYELONEPHRITIS CHRONIC (Infections and infestations) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RED BLOOD CELL COUNT INCREASED (Investigations) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 6 (6) | 6 (6)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
RESPIRATORY FUME INHALATION DISORDER (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RESPIRATORY GAS EXCHANGE DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (5) | 3 (3)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (2)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 34 (42) | 41 (49)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
RUPTURED ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
SALPINGECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
SARCOIDOSIS (Immune system disorders) | 1 (1) | 0 (0)
SCHIZOAFFECTIVE DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
SCLERODERMA ASSOCIATED DIGITAL ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
SECONDARY IMMUNODEFICIENCY (Immune system disorders) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 3 (3) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 3 (3) | 1 (1)
SIGMOIDITIS (Gastrointestinal disorders) | 0 (0) | 1 (2)
SKIN NEOPLASM EXCISION (Surgical and medical procedures) | 1 (2) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SOMNAMBULISM (Psychiatric disorders) | 0 (0) | 1 (1)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
STEM CELL TRANSPLANT (Surgical and medical procedures) | 1 (2) | 0 (0)
STILL'S DISEASE ADULT ONSET (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
STRESS (Psychiatric disorders) | 1 (1) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
SUDDEN CARDIAC DEATH (General disorders) | 1 (1) | 0 (0)
SUDDEN DEATH (General disorders) | 5 (5) | 4 (4)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 4 (6)
SYNCOPE (Nervous system disorders) | 10 (13) | 20 (23)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
SYSTEMIC SCLEROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
TACHYCARDIA (Cardiac disorders) | 1 (2) | 0 (0)
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
THALAMIC INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TRACHEOBRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 (2) | 0 (0)
TRANSPLANT EVALUATION (Investigations) | 1 (1) | 0 (0)
TRAUMATIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TURBINECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (3) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 3 (3)
URETHRAL OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0)
URETHRAL STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
VACCINATION COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 2 (2) | 0 (0)
VENA CAVA THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
VENOUS INSUFFICIENCY (Vascular disorders) | 0 (0) | 1 (1)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 3 (3) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2)
WALKING DISTANCE TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selexipag (N=575) | Placebo (N=577)
ABDOMINAL PAIN (Gastrointestinal disorders) | 44 (54) | 29 (37)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 34 (39) | 32 (38)
ANAEMIA (Blood and lymphatic system disorders) | 43 (53) | 28 (37)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 62 (82) | 44 (57)
ASTHENIA (General disorders) | 29 (33) | 24 (27)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 34 (36) | 35 (38)
BRONCHITIS (Infections and infestations) | 42 (46) | 41 (49)
CHEST PAIN (General disorders) | 34 (37) | 39 (54)
COUGH (Respiratory, thoracic and mediastinal disorders) | 56 (67) | 67 (87)
DECREASED APPETITE (Metabolism and nutrition disorders) | 34 (38) | 19 (23)
DIARRHOEA (Gastrointestinal disorders) | 242 (375) | 109 (137)
DIZZINESS (Nervous system disorders) | 85 (111) | 85 (106)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 79 (100) | 110 (143)
FATIGUE (General disorders) | 46 (54) | 58 (72)
FLUSHING (Vascular disorders) | 69 (80) | 29 (31)
HEADACHE (Nervous system disorders) | 374 (649) | 189 (261)
MYALGIA (Musculoskeletal and connective tissue disorders) | 90 (120) | 34 (37)
NASOPHARYNGITIS (Infections and infestations) | 75 (105) | 63 (95)
NAUSEA (Gastrointestinal disorders) | 192 (265) | 107 (136)
OEDEMA PERIPHERAL (General disorders) | 77 (90) | 100 (138)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 95 (142) | 46 (62)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 148 (188) | 36 (38)
PALPITATIONS (Cardiac disorders) | 32 (40) | 31 (41)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 46 (64) | 84 (141)
SYNCOPE (Nervous system disorders) | 30 (35) | 34 (42)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 72 (100) | 79 (119)
URINARY TRACT INFECTION (Infections and infestations) | 24 (30) | 30 (34)
VOMITING (Gastrointestinal disorders) | 103 (143) | 48 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less